CLINICAL TRIAL: NCT04905784
Title: The Impact of Simple Home-based Differential Learning on Oral Hygiene in Children: A Single-blind Randomized Controlled Clinical Trial
Brief Title: The Impact of Simple Home-based Differential Learning on Oral Hygiene in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZZMK KiZHK BB 031/21
Record Dates: First submitted 2021-05-03; First posted 2021-05-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Dental Caries; Gingival Diseases
Keywords: Caries; Dental; Prevention; Differential; Learning; Toothbrushing
MeSH Terms: conditions — Dental Caries; Gingival Diseases

STUDY DESIGN:
Intervention Model Description: Parallel group, single-blind randomized controlled clinical trial.
Who Masked: Investigator
Masking Description: The information and instructions for the two groups will be placed in 70 envelopes, each group has 35 envelopes, and then these envelopes will be mixed randomly (as in playing cards) and at the end these envelopes will be placed in a box. Patients will be asked to randomly select an envelope from the box. The investigator assesses oral hygiene in check-up appointments without knowledge of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Usual brushing. (Active Comparator): Usual motivation to brush teeth in the clinic (KAI brushing technique) in addition to brushing teeth by the parents.
  Interventions: Behavioral: Usual toothbrushing
- Test group: Differential learning group. (Experimental): Use of differential learning of tooth brushing at home, including children and parents.
  Interventions: Behavioral: Differential learning

INTERVENTIONS:
Behavioral: Differential learning — The patient will be requested to perform different exercises, each exercise one time a day for 3 days in a row before moving to the next exercise. All patient will be asked to do the exercises in the same sequence.
  Arms: Test group: Differential learning group.
Behavioral: Usual toothbrushing — The patients in this group will be provided with the regular oral health instructions, including the traditional toothbrushing recommendations.
  Arms: Control group: Usual brushing.

SUMMARY:
This randomized clinical trial study aims to investigate the impact of home-based differential learning on tooth brushing, in particular on the reduction of plaque and maintenance of gingival health in children aged 3 to 8 years, compared to the habitual tooth brushing and instruction/demonstration tooth brushing learning method.

DETAILED DESCRIPTION:
This two-parallel arm single-blind randomized controlled clinical trial will be undertaken at the Department of Preventive and Pediatric Dentistry at the University of Greifswald. The examination of the patient will be undertaken in a dental chair set up using standard infection control guidelines for a dental examination used at the department. The allocation of the patients to the two groups will be done through asking the patients to pick up an envelope randomly from a box which contains the information and explanation for home brushing.

In the first visit, the baseline dental examination and patient acceptance survey will be done to comprehensively assess each participant's oral health status, their oral hygiene status, caries experience and periodontal condition will be recorded.

To assess oral hygiene status we will use plaque index (PI) (Quigley Hein, 1972) on a scale of 0 to 5. Dental caries experience will be recorded by counting the numbers of teeth that are decayed (dt/DT), missing due to caries (mt/MT), and filled (ft/FT) to generate a dmft/DMFT score. Periodontal condition will be recorded using the papillary bleeding index Index (PBI) on a scale of 0 to 4. One trained and calibrated examiner will perform the clinical examinations.

The study and its objectives will be explained to the patients. For the control group, regular instructions and advice will be provided as in any regular prophylaxis session.

For the test group, the exercises and movements to be performed when brushing the teeth will be explained. The patients in both groups will be also provided with explanation leaflet with the exercises and a free toothbrush. There will be no restriction on the type of the fluoridated toothpaste.

The training sheet will include the following exercises:

* Tooth brushing while lying down.
* Tooth brushing with one eye covered (i.e. with the hand).
* Tooth brushing wearing large gloves.
* Tooth brushing with the non-dominant hand.
* Tooth brushing using both hands.
* Different sequence of tooth brushing compared to the practical demonstration (i.e. starting with cleaning the lingual surface instead of occlusal surface).
* Tooth brushing while both eyes are closed.
* Tooth brushing with an obstruction on the elbow of the dominant hand (i.e. wraps a piece of cloth/ scarf around the elbow).
* Tooth brushing while watching 3-5 minutes video (i.e. using YouTube). The parent/ child will be requested to perform each exercise one time a day for 3 days in a row before moving to the next exercise. All parent/ child will be asked to do the exercises in the same sequence. After completing the exercise for each day, children will be asked to put a sticker in the calendar table, which will be provided to them as a motivation to perform the exercises.

There will be 2 follow-ups; the first follow-up after one month will include dental re-examination, using the same methods and criteria as the baseline examination as well as a questionnaire for the parents to assess their experience and acceptance of the used method. The second follow-up will be after 3 months and it will include dental re-examination, using the same methods and criteria as the baseline examination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 - 8 years.
* Need for parental assistance with tooth brushing.
* Need for check-up/ prophylaxis appointment approx. 4 and 12 weeks.

Exclusion Criteria:

* Patients with pain/ patients with signs or symptoms to be treated.
* Patients with systemic disease that require special attention during their dental treatment.
* Parents / children who refuse to participate in the study.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Oral hygiene - dental plaque | 1 month
  Plaque index (QHI: Quigley-Hein plaque index)
Oral hygiene - dental plaque | 3 months
  Plaque index (QHI: Quigley-Hein plaque index)
Oral hygiene - gingivitis | 1 month
  Gingival bleeding index (PBI: papilla bleeding index)
Oral hygiene - gingivitis | 3 months
  Gingival bleeding index (PBI: papilla bleeding index)

SECONDARY OUTCOMES:
Parental acceptance | 1 month
  self-designed questionnaire about the acceptance (11 items), assessment using five-point Likert-scale which is from 1 (minimal value) to 5 (maximal value) e.g. with 5 strongly agree and 1 strongly disagree
Parental acceptance (mid-term) | 3 months
  self-designed questionnaire about the acceptance (11 items), assessment using five-point Likert-scale which is from 1 (minimal value) to 5 (maximal value) e.g. with 5 strongly agree and 1 strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Loay Leghrouz, M.Sc., Principal Investigator — Universitätmedizin Greifswald
Locations (2):
- Germany (2):
  - Universitätmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - University medicine Greifswald, Greifswald

IPD SHARING:
Plan to Share IPD: No